CLINICAL TRIAL: NCT01683266
Title: A 6-Month, Multicenter, Randomized, Open-label, Parallel-group Study Comparing the Efficacy and Safety of a New Formulation of Insulin Glargine and Lantus® Injected in the Morning or Evening in Patients With Type 1 Diabetes Mellitus With a 6-month Safety Extension Period
Brief Title: Comparison of a New Formulation of Insulin Glargine With Lantus in Patients With Type 1 Diabetes Mellitus
Acronym: EDITION IV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC12456; 2012-001524-35 (EudraCT Number); U1111-1128-5517 (Other: UTN)
Record Dates: First submitted 2012-09-07; First posted 2012-09-11 (Estimated); Results first posted 2015-04-23 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-05

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HOE901-U300 (Experimental): HOE901-U300 (new insulin glargine 300 units per milliliter [U/mL]) subcutaneous (SC) injection once daily in morning or evening for 12 months on top of mealtime insulin analogue. Dose titration seeking fasting plasma glucose 4.4-5.6 millimole per liter (mmol/L) (80 - 100 milligram per deciliter [mg/dL]).
  Interventions: Drug: HOE901-U300 (Insulin glargine new formulation)
- Lantus (Active Comparator): Lantus (HOE901-U100, insulin glargine 100 U/mL) SC injection once daily in morning or evening for 12 months on top of mealtime insulin analogue. Dose titration seeking fasting plasma glucose 4.4-5.6 mmol/L (80 - 100 mg/dL).
  Interventions: Drug: Lantus (Insulin glargine)

INTERVENTIONS:
Drug: HOE901-U300 (Insulin glargine new formulation)
  Arms: HOE901-U300
Drug: Lantus (Insulin glargine)
  Arms: Lantus

SUMMARY:
Primary Objective:

* To compare the efficacy of a new formulation of insulin glargine and Lantus (overall, regardless the injection time) in terms of change of HbA1c from baseline to endpoint (scheduled Month 6) in participants with type 1 diabetes mellitus

Secondary Objective:

* To compare HOE901-U300 and Lantus when given in the morning or in the evening in terms of:
* Change of HbA1c from baseline to endpoint (scheduled Month 6)
* Change from baseline to endpoint (Month 6) in fasting plasma glucose (FPG), plasma glucose prior to injection of study drug, plasma glucose at 03:00 hours, mean plasma glucose (8-point profiles), glucose variability, treatment satisfaction and health related quality of life in participants with Type 1 Diabetes Mellitus (T1DM)
* Reaching target HbA1c values and controlled plasma glucose (all and reaching target without hypoglycemia)
* Frequency of occurrence and diurnal distribution of hypoglycemia by category of hypoglycemia (symptomatic, asymptomatic, nocturnal, severe, probable and relative)
* Safety and tolerability of HOE901-U300 including development of anti-insulin antibody (AIAs) during the 12-month study period

DETAILED DESCRIPTION:
The maximum study duration was up to approximately 54 weeks per participants:

* Up to 2-week screening period
* 6-month open-label comparative efficacy and safety treatment period
* 6-month open-label comparative safety extension period
* 48-hour post-treatment safety follow-up period

ELIGIBILITY:
Inclusion criteria:

* Adult participants with type 1 diabetes mellitus

Exclusion criteria:

* HbA1c less than (<) 7.0% (53 mmol/mol) or greater than (>) 10% (86 mmol/mol) at screening
* Less than 1 year on any basal plus mealtime insulin and self-monitoring of blood glucose before screening visit
* Participants not on stable insulin dose (+/-20 percent total basal insulin dose) in the last 30 days prior to screening visit
* Participants using pre-mix insulins, human regular insulin as mealtime insulin and/or any glucose-lowering drugs other than basal insulin and mealtime analogue insulin in the last 3 months before screening visit
* Use of an insulin pump in the last 6 months before screening visit and no plan to switch to insulin pump in the next 12 months
* Not willing to inject insulin glargine as assigned by the randomization process once daily in the morning or evening;
* Severe hypoglycemia resulting in coma/seizures, and/or hospitalization for diabetic ketoacidosis in the last 6 months before screening visit
* Unstable proliferative diabetic retinopathy or any other rapidly progressive diabetic retinopathy or macular edema likely to require treatment (example laser, surgical treatment or injectable drugs) during the study period

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 549 (Actual)
Dates: Start 2012-09; Primary Completion 2013-09 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (147):
- United States (82):
  - Investigational Site Number 840156, Chandler, Arizona
  - Investigational Site Number 840177, Little Rock, Arkansas
  - Investigational Site Number 840430, Bell Gardens, California
  - Investigational Site Number 840131, Escondido, California
  - Investigational Site Number 840140, Fresno, California
  - Investigational Site Number 840107, Greenbrae, California
  - Investigational Site Number 840149, Huntington Beach, California
  - Investigational Site Number 840120, La Jolla, California
  - Investigational Site Number 840123, La Mesa, California
  - Investigational Site Number 840159, La Mesa, California
  - Investigational Site Number 840114, Long Beach, California
  - Investigational Site Number 840189, Mission Hills, California
  - Investigational Site Number 840105, Temecula, California
  - Investigational Site Number 840155, Tustin, California
  - Investigational Site Number 840115, Walnut Creek, California
  - Investigational Site Number 840160, Denver, Colorado
  - Investigational Site Number 840188, Denver, Colorado
  - Investigational Site Number 840196, New Haven, Connecticut
  - Investigational Site Number 840113, Bradenton, Florida
  - Investigational Site Number 840102, Hialeah, Florida
  - Investigational Site Number 840134, Hollywood, Florida
  - Investigational Site Number 840185, Jacksonville, Florida
  - Investigational Site Number 840116, Jacksonville, Florida
  - Investigational Site Number 840126, Miami, Florida
  - Investigational Site Number 840179, Miami, Florida
  - Investigational Site Number 840117, New Port Richey, Florida
  - Investigational Site Number 840174, Orlando, Florida
  - Investigational Site Number 840110, Oviedo, Florida
  - Investigational Site Number 840178, Palm Harbor, Florida
  - Investigational Site Number 840181, Tampa, Florida
  - Investigational Site Number 840420, West Palm Beach, Florida
  - Investigational Site Number 840195, Atlanta, Georgia
  - Investigational Site Number 840124, Honolulu, Hawaii
  - Investigational Site Number 840167, Idaho Falls, Idaho
  - Investigational Site Number 840163, Nampa, Idaho
  - Investigational Site Number 840162, Springfield, Illinois
  - Investigational Site Number 840172, Avon, Indiana
  - Investigational Site Number 840197, Indianapolis, Indiana
  - Investigational Site Number 840108, Des Moines, Iowa
  - Investigational Site Number 840407, Iowa City, Iowa
  - Investigational Site Number 840170, Topeka, Kansas
  - Investigational Site Number 840421, Lexington, Kentucky
  - Investigational Site Number 840426, Metairie, Louisiana
  - Investigational Site Number 840104, Baltimore, Maryland
  - Investigational Site Number 840180, Rockville, Maryland
  - Investigational Site Number 840137, Haverhill, Massachusetts
  - Investigational Site Number 840408, Detroit, Michigan
  - Investigational Site Number 840153, Madison Heights, Michigan
  - Investigational Site Number 840171, Saint Louis Park, Minnesota
  - Investigational Site Number 840184, St Louis, Missouri
  - Investigational Site Number 840106, Omaha, Nebraska
  - Investigational Site Number 840145, Omaha, Nebraska
  - Investigational Site Number 840139, Las Vegas, Nevada
  - Investigational Site Number 840151, Albuquerque, New Mexico
  - Investigational Site Number 840191, New Hyde Park, New York
  - Investigational Site Number 840173, Syracuse, New York
  - Investigational Site Number 840133, Asheville, North Carolina
  - Investigational Site Number 840175, Chapel Hill, North Carolina
  - Investigational Site Number 840161, Morganton, North Carolina
  - Investigational Site Number 840169, Mentor, Ohio
  - Investigational Site Number 840119, Norman, Oklahoma
  - Investigational Site Number 840112, Bend, Oregon
  - Investigational Site Number 840136, Greer, South Carolina
  - Investigational Site Number 840122, Dakota Dunes, South Dakota
  - Investigational Site Number 840144, Chattanooga, Tennessee
  - Investigational Site Number 840187, Nashville, Tennessee
  - Investigational Site Number 840109, Austin, Texas
  - Investigational Site Number 840157, Austin, Texas
  - Investigational Site Number 840150, Dallas, Texas
  - Investigational Site Number 840412, Dallas, Texas
  - Investigational Site Number 840130, Houston, Texas
  - Investigational Site Number 840141, Houston, Texas
  - Investigational Site Number 840166, San Antonio, Texas
  - Investigational Site Number 840101, Murray, Utah
  - Investigational Site Number 840125, Burke, Virginia
  - Investigational Site Number 840427, Chesapeake, Virginia
  - Investigational Site Number 840103, Manassas, Virginia
  - Investigational Site Number 840132, Renton, Washington
  - Investigational Site Number 840403, Seattle, Washington
  - Investigational Site Number 840402, Spokane, Washington
  - Investigational Site Number 840127, Tacoma, Washington
  - Investigational Site Number 840411, Milwaukee, Wisconsin
- Canada (6):
  - Investigational Site Number 124110, Coquitlam
  - Investigational Site Number 124104, Laval
  - Investigational Site Number 124108, Mirabel
  - Investigational Site Number 124109, Montreal
  - Investigational Site Number 124105, Thornhill
  - Investigational Site Number 124101, Toronto
- Czechia (3):
  - Investigational Site Number 203102, Brno
  - Investigational Site Number 203104, Prague
  - Investigational Site Number 203103, Prague
- Denmark (5):
  - Investigational Site Number 208102, Aalborg
  - Investigational Site Number 208103, Esbjerg
  - Investigational Site Number 208105, Gentofte Municipality
  - Investigational Site Number 208104, København NV
  - Investigational Site Number 208107, Køge
- Estonia (5):
  - Investigational Site Number 233104, Pärnu
  - Investigational Site Number 233105, Tallinn
  - Investigational Site Number 233106, Tartu
  - Investigational Site Number 233101, Tartu
  - Investigational Site Number 233103, Viljandimaa
- Finland (5):
  - Investigational Site Number 246102, Kokkola
  - Investigational Site Number 246101, Kuopio
  - Investigational Site Number 246106, Loimaa
  - Investigational Site Number 246105, Oulu
  - Investigational Site Number 246103, Tampere
- Hungary (6):
  - Investigational Site Number 348103, Budapest
  - Investigational Site Number 348108, Budapest
  - Investigational Site Number 348107, Budapest
  - Investigational Site Number 348106, Debrecen
  - Investigational Site Number 348102, Gyula
  - Investigational Site Number 348101, Úrhida
- Japan (11):
  - Investigational Site Number 392110, Aisai
  - Investigational Site Number 392105, Ise-Shi
  - Investigational Site Number 392104, Karatsu-Shi
  - Investigational Site Number 392111, Kitakyushu-Shi
  - Investigational Site Number 392108, Matsumoto
  - Investigational Site Number 392112, Matsumoto-Shi
  - Investigational Site Number 392103, Midori
  - Investigational Site Number 392107, Mito
  - Investigational Site Number 392101, Sakaishi
  - Investigational Site Number 392102, Tomishiro
  - Investigational Site Number 392106, Yamagata
- Latvia (5):
  - Investigational Site Number 428106, Limbaži
  - Investigational Site Number 428103, Riga
  - Investigational Site Number 428105, Riga
  - Investigational Site Number 428102, Sigulda
  - Investigational Site Number 428101, Ventspils
- Netherlands (5):
  - Investigational Site Number 528101, Almere Stad
  - Investigational Site Number 528103, Beek
  - Investigational Site Number 528105, Nijmegen
  - Investigational Site Number 528104, Venlo
  - Investigational Site Number 528102, Zwijndrecht
- Investigational Site Number 840602, Ponce, Puerto Rico
- Romania (9):
  - Investigational Site Number 642107, Bacau
  - Investigational Site Number 642103, Brasov
  - Investigational Site Number 642109, Oradea
  - Investigational Site Number 642106, Reşiţa
  - Investigational Site Number 642104, Sibiu
  - Investigational Site Number 642101, Târgu Mureş
  - Investigational Site Number 642102, Târgu Mureş
  - Investigational Site Number 642105, Timișoara
  - Investigational Site Number 642108, Timișoara
- Sweden (4):
  - Investigational Site Number 752103, Gothenburg
  - Investigational Site Number 752105, Kristianstad
  - Investigational Site Number 752101, Stockholm
  - Investigational Site Number 752104, Vällingby

REFERENCES:
- [Derived] Home PD, Bergenstal RM, Bolli GB, Ziemen M, Rojeski M, Espinasse M, Riddle MC. Glycaemic control and hypoglycaemia during 12 months of randomized treatment with insulin glargine 300 U/mL versus glargine 100 U/mL in people with type 1 diabetes (EDITION 4). Diabetes Obes Metab. 2018 Jan;20(1):121-128. doi: 10.1111/dom.13048. Epub 2017 Aug 8. PMID 28661585

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 846 participants were screened, of whom 297 participants were screen failure and 549 participants were randomized.
Groups:
- HOE901--U300: HOE901-U300 (new insulin glargine 300 units per milliliter [U/mL]) subcutaneous (SC) injection once daily in morning or evening for 12 months on top of mealtime insulin analogue.
- Lantus: Lantus (HOE901-U100, insulin glargine 100 U/mL) SC injection once daily in morning or evening for 12 months on top of mealtime insulin analogue.
Period: Overall Study
Arm/Group | HOE901--U300 | Lantus
Started | 274 | 275
Modified Intent-to-Treat Population | 273 (Participants who received at least 1 dose of drug, had both baseline, at least 1 post-baseline data) | 273 (Participants who received at least 1 dose of drug, had both baseline, at least 1 post-baseline data)
Completed | 219 | 225
Not Completed | 55 | 50
Not completed — Adverse Event | 5 | 4
Not completed — Lack of Efficacy | 5 | 2
Not completed — Protocol Violation | 13 | 6
Not completed — Personal Reason | 17 | 25
Not completed — Selection Criterion / Protocol Violation | 7 | 5
Not completed — Lost to Follow-up | 5 | 0
Not completed — Site Closure / Site Withdrawal | 1 | 3
Not completed — Nonserious Hypoglycemia | 0 | 3
Not completed — Perceived Lack of Efficacy | 1 | 1
Not completed — Possibly Hypoglycemia | 1 | 0
Not completed — Serious Adverse Event of Hypoglycemia | 0 | 1

BASELINE CHARACTERISTICS:
Population: Randomized population: all screened participants (who originally met inclusion criteria and signed informed consent) allocated to a treatment group and recorded in Interactive Voice/Web Response System (IVRS/IWRS) database, regardless of whether treatment was used or not. Participants were analyzed in treatment group to which they were randomized.
Groups:
- HOE901--U300: HOE901-U300 SC injection once daily in morning or evening for 12 months on top of mealtime insulin.
- Lantus: Lantus SC injection once daily in morning or evening for 12 months on top of mealtime insulin.
- Total: Total of all reporting groups
Arm/Group | HOE901--U300 | Lantus | Total
Number analyzed (Participants) | 274 | 275 | 549
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (13.9) | 48.2 (13.4) | 47.3 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 111 | 236
  Male | 149 | 164 | 313
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 27.6 (5.5) | 27.6 (4.7) | 27.6 (5.1)
Duration of Diabetes [Mean (Standard Deviation); unit: years] — Number of participants analyzed for this baseline characteristics = 274 and 272 for each reporting group, respectively.
  years | 20.5 (12.7) | 21.4 (13.1) | 21.0 (12.9)
Glycated Hemoglobin (HbA1c) [Number; unit: participants]
  Less Than (<) 8% | 105 | 105 | 210
  Greater Than or Equal to (>=) 8% | 169 | 170 | 339
Basal Insulin Daily Dose [Mean (Standard Deviation); unit: units per kilogram (U/kg)] — Number of participants analyzed for this baseline characteristics = 201 and 210 for each reporting group, respectively.
  units per kilogram (U/kg) | 0.381 (0.173) | 0.372 (0.152) | 0.376 (0.162)
Total Insulin Daily Dose [Mean (Standard Deviation); unit: U/kg] — Number of participants analyzed for this baseline characteristics = 195 and 198 for each reporting group, respectively.
  U/kg | 0.714 (0.278) | 0.724 (0.245) | 0.719 (0.262)

OUTCOME MEASURES:

1. Primary Outcome: Change In HbA1c From Baseline to Month 6 Endpoint
Time Frame: Baseline, Month 6
Population: Modified Intent-to-Treat (mITT) population: all randomized participants who received at least (>=)1 dose, had baseline and >=1 post-baseline assessment of any efficacy variable, irrespective of compliance. Number of participants analyzed = participants with baseline and Month 6 HbA1c assessment.
Measure: Least Squares Mean (Standard Error); unit: percentage of hemoglobin
Arm/Group | HOE901--U300 | Lantus
Number analyzed (Participants) | 225 | 229
percentage of hemoglobin | -0.40 (0.051) | -0.44 (0.051)
Statistical Analysis 1: Comparison: HOE901--U300 vs Lantus; Analysis was performed using mixed model for repeated measurements (MMRM) with treatment groups, strata of screening HbA1c (<8.0, >=8.0%), geographical region (Non-Japan; Japan), visit and visit-by-treatment groups interaction as fixed categorical effects; baseline HbA1c and baseline HbA1c-by-visit interaction as continuous fixed covariates; Test type: Non-Inferiority or Equivalence — Stepwise closed testing approach was used to assess non-inferiority and superiority sequentially: 1. Non-inferiority of HOE901-U300 vs Lantus: Upper bound of two-sided 95% confidence interval (CI) of difference between HOE901-U300 and Lantus on mITT population is <0.4%. 2. Superiority (only if non-inferiority has been demonstrated): Upper bound of two-sided 95% CI for difference in mean change in HbA1c from baseline to endpoint between HOE901-U300 and Lantus on mITT population is <0; Least Squares (LS) Mean difference = 0.04, 95% CI 2-sided [-0.098 to 0.185], Standard Error of Mean 0.072

2. Secondary Outcome: Percentage of Participants With HbA1c <7% at Month 6 Endpoint
Time Frame: Month 6
Population: mITT Population.
Measure: Number; unit: percentage of participants
Arm/Group | HOE901--U300 | Lantus
Number analyzed (Participants) | 273 | 273
percentage of participants | 16.8 | 15.0

3. Secondary Outcome: Percentage of Participants With HbA1c Less Than or Equal to 6.5% at Month 6 Endpoint
Time Frame: Month 6
Population: mITT Population.
Measure: Number; unit: percentage of participants
Arm/Group | HOE901--U300 | Lantus
Number analyzed (Participants) | 273 | 273
percentage of participants | 8.1 | 5.5

4. Secondary Outcome: Change In Average Pre-Injection Self-Monitored Plasma Glucose (SMPG) From Baseline Month 6 Endpoint
Description: Pre-injection SMPG was measured within 30 minutes prior to the injection of the study drug. Average was assessed by the mean of at least 3 SMPG calculated over the 7 days preceding the assessment visit.
Time Frame: Baseline, Month 6
Population: mITT population. Number of participants analyzed = participants with baseline and Month 6 pre-injection SMPG assessment.
Measure: Least Squares Mean (Standard Error); unit: millimole per liter (mmol/L)
Arm/Group | HOE901--U300 | Lantus
Number analyzed (Participants) | 117 | 105
millimole per liter (mmol/L) | -1.16 (0.223) | -0.82 (0.233)
Statistical Analysis 1: Comparison: HOE901--U300 vs Lantus; Change in pre-injection SMPG was analyzed using MMRM model with treatment groups, strata of screening HbA1c (<8.0, >=8.0%), geographical region (Non-Japan; Japan), visit and visit-by-treatment groups interaction as fixed categorical effects; pre-injection SMPG value and pre-injection SMPG value-by-visit interaction as continuous fixed covariates; Test type: Superiority or Other; LS Mean difference = -0.35, 95% CI 2-sided [-0.982 to 0.287], Standard Error of Mean 0.322

5. Secondary Outcome: Change in Variability of Pre-injection SMPG From Baseline to Month 6 Endpoint
Description: Pre-injection SMPG was measured within 30 minutes prior to the injection of the study drug. Variability was assessed by the mean of coefficient of variation calculated as 100 multiplied by (standard deviation/mean) over at least 3 SMPG measured during the 7 days preceding the assessment visit.
Time Frame: Baseline, Month 6
Population: mITT population. Number of participants analyzed = participants with baseline and Month 6 pre-injection SMPG assessment.
Measure: Least Squares Mean (Standard Error); unit: percentage of mean
Arm/Group | HOE901--U300 | Lantus
Number analyzed (Participants) | 117 | 105
percentage of mean | -3.03 (1.573) | -1.76 (1.651)

6. Secondary Outcome: Change in Fasting Plasma Glucose From Baseline to Month 6 Endpoint
Time Frame: Baseline, Month 6
Population: mITT Population. Number of participants analyzed = participants with baseline and Month 6 FPG assessment.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | HOE901--U300 | Lantus
Number analyzed (Participants) | 213 | 216
mmol/L | -0.95 (0.263) | -1.14 (0.260)

7. Secondary Outcome: Percentage of Participants With Fasting Plasma Glucose (FPG) <5.6 mmol/L (100 mg/dL) At Month 6
Time Frame: Month 6
Population: mITT Population.
Measure: Number; unit: percentage of participants
Arm/Group | HOE901--U300 | Lantus
Number analyzed (Participants) | 273 | 273
percentage of participants | 9.9 | 12.8

8. Secondary Outcome: Percentage of Participants With FPG <7.2 mmol/L (130 mg/dL) at Month 6 Endpoint
Time Frame: Month 6
Population: mITT Population. Number of participants analyzed = participants with baseline and Month 6 FPG assessment.
Measure: Number; unit: percentage of participants
Arm/Group | HOE901--U300 | Lantus
Number analyzed (Participants) | 273 | 273
percentage of participants | 25.3 | 25.6

9. Secondary Outcome: Change in 8--Point SMPG Profiles Per Time Point From Baseline to Month 6 Endpoint
Description: Change in each time-point of 8-point SMPG profile: 03:00 hours (clock time) at night; before and 2 hours after breakfast; before and 2 hours after lunch; before and 2 hours after dinner; and at bedtime.
Time Frame: Baseline, Month 6
Population: mITT Population. Here, n = participants with Baseline and Month 6 8-point SMPG assessment separately for each analysed time point.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | HOE901--U300 | Lantus
Number analyzed (Participants) | 273 | 273
mmol/L
  03:00 at Night (n= 156, 159) | -0.47 (4.56) | -0.67 (4.98)
  Pre--Breakfast (n= 166, 167) | -0.86 (5.30) | -0.07 (5.20)
  2 Hours After Breakfast (n= 152, 156) | -0.62 (4.75) | -1.18 (5.66)
  Pre--Lunch (n= 166, 166) | -0.95 (4.53) | -0.93 (4.76)
  2 Hours After Lunch (n= 163,163) | -0.13 (5.20) | -1.43 (5.37)
  Pre--Dinner (n= 165,166) | -0.56 (6.00) | -1.74 (5.28)
  2 Hours After Dinner (n= 154,152) | -0.93 (5.27) | -1.19 (5.51)
  Bedtime (n= 141,146) | -0.80 (5.39) | -1.91 (5.10)

10. Secondary Outcome: Change in Daily Average Total Insulin Dose From Baseline to Month 6 Endpoint
Time Frame: Baseline, Month 6
Population: mITT Population. Number of participants analyzed = participants with Baseline and Month 6 daily average total insulin dose assessment.
Measure: Mean (Standard Deviation); unit: U/kg
Arm/Group | HOE901--U300 | Lantus
Number analyzed (Participants) | 173 | 158
U/kg | 0.19 (0.22) | 0.10 (0.16)

11. Secondary Outcome: Change in Total Treatment Satisfaction Score Using The Diabetes Treatment Satisfaction Questionnaire (DTSQs) From Baseline to Month 6 Endpoint
Description: DTSQ is a validated measure to assess how satisfied participants with diabetes are with their treatment and how they perceive hyper- and hypoglycemia. It consists of 8 questions which are answered on a Likert scale from 0 to 6. DTSQ treatment satisfaction score is the sum of question 1 and 4-8 scores and ranges between 0 and 36, where higher scores indicate more treatment satisfaction.
Time Frame: Baseline, Month 6
Population: mITT Population. Number of participants analyzed = participants with Baseline and Month 6 DTSQ assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | HOE901--U300 | Lantus
Number analyzed (Participants) | 212 | 206
units on a scale | 1.00 (0.331) | 1.41 (0.334)

12. Secondary Outcome: Percentage of Participants With Hypoglycemia (All and Nocturnal) Events From Baseline to Month 12
Description: Hypoglycemia events were Severe hypoglycemia (an event that required assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions); Documented symptomatic hypoglycemia (typical symptoms of hypoglycemia with plasma glucose level of <=3.9 mmol/L [70 mg/dL]); Asymptomatic hypoglycemia (no typical symptoms of hypoglycemia but plasma glucose level <=3.9 mmol/L); Probable symptomatic hypoglycemia (an event during which symptoms of hypoglycemia were not accompanied by a plasma glucose determination, but was presumably caused by a plasma glucose level <=3.9 mmol/L, symptoms treated with oral carbohydrate without a test of plasma glucose); Relative hypoglycemia (an event during which the person with diabetes reported any of the typical symptoms of hypoglycemia, and interpreted the symptoms as indicative of hypoglycemia, but plasma glucose level >3.9 mmol/L); Severe and/or confirmed a hypoglycemia (plasma glucose <=3.9 mmol/L).
Time Frame: Up to Month 12
Population: Safety population: all participants randomized and exposed to at least one dose of study drug, regardless of the amount of treatment administered. In the event of participants having received treatments different from those assigned according to the randomization schedule, safety analyses were conducted according to treatment received.
Measure: Number; unit: percentage of participants
Arm/Group | HOE901--U300 | Lantus
Number analyzed (Participants) | 274 | 275
percentage of participants
  Any Hypoglycemia Event: All Hypoglycemia | 95.3 | 94.9
  Severe Hypoglycemia: All Hypoglycemia | 9.1 | 11.3
  Documented Symptomatic: All Hypoglycemia | 87.6 | 86.5
  Asymptomatic: All Hypoglycemia | 76.6 | 81.5
  Probable Symptomatic: All Hypoglycemia | 11.3 | 15.3
  Relative: All Hypoglycemia | 14.6 | 9.5
  Severe and/or Confirmed: All Hypoglycemia | 94.9 | 94.5
  Any Hypoglycemia Event: Nocturnal Hypoglycemia | 73.4 | 74.9
  Severe Hypoglycemia: Nocturnal Hypoglycemia | 3.3 | 3.3
  Documented Symptomatic: Nocturnal Hypoglycemia | 64.2 | 63.3
  Asymptomatic: Nocturnal Hypoglycemia | 35.0 | 38.9
  Probable Symptomatic: Nocturnal Hypoglycemia | 5.1 | 6.5
  Relative: Nocturnal Hypoglycemia | 4.0 | 5.5
  Severe and/or Confirmed: Nocturnal Hypoglycemia | 72.6 | 74.5

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of informed consent form up to study completion regardless of seriousness or relationship to study drug.
Description: Reported adverse events are treatment-emergent adverse events that is AEs that developed/worsened during the 'on treatment period' (as the time from first injection of IMP up to 2 days after the last injection of IMP). Analysis was done on safety population.
Arm/Group | HOE901--U300 | Lantus
Serious Adverse Events (participants affected / at risk) | 27/274 | 26/275
Other Adverse Events (participants affected / at risk) | 113/274 | 86/275
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HOE901--U300 (N=274) | Lantus (N=275)
Angina pectoris (Cardiac disorders) | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Chronic tonsillitis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0
H1N1 influenza (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Brain contusion (Injury, poisoning and procedural complications) | 0 | 1
Comminuted fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Open fracture (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 16 | 13
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Aphasia (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0
Diabetic neuropathy (Nervous system disorders) | 0 | 1
Hypoglycaemic seizure (Nervous system disorders) | 1 | 1
Hypoglycaemic unconsciousness (Nervous system disorders) | 1 | 1
Loss of consciousness (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Femoral artery occlusion (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HOE901--U300 (N=274) | Lantus (N=275)
Influenza (Infections and infestations) | 16 | 14
Nasopharyngitis (Infections and infestations) | 43 | 35
Sinusitis (Infections and infestations) | 14 | 11
Upper respiratory tract infection (Infections and infestations) | 38 | 26
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 7
Headache (Nervous system disorders) | 17 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.